CLINICAL TRIAL: NCT05897398
Title: SEMASEARCH, Retrospective/Prospective Cohort Nested at ATUc/AP2 WEGOVY®
Acronym: SEMASEARCH
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0954
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Bariatric Surgery; Binge Eating Disorder; Syndromic Obesity; Sarcopenic Obesity; Iatrogenic Obesity; Psychotropic Drugs
Keywords: Obesity; Semaglutide; WEGOVY®
MeSH Terms: conditions — Obesity; Binge-Eating Disorder | interventions — Data Collection; Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients already receiving WEGOVY® treatment included in the ATUc/AP2: Data collected at initiation, 6 months and 12 months of WEGOVY® treatment will be retrospectively extracted from the WEGOVY® ATU/AP2 eCRF.
  Interventions: Other: Data collection; Other: Blood sampling; Other: Questionnaires

INTERVENTIONS:
Other: Data collection — Data collected at initiation, 6 months and 12 months of WEGOVY® treatment will be retrospectively extracted from the WEGOVY® ATU/AP2 eCRF.
Other: Blood sampling — Blood sampling for routine care (max 15mL)
Other: Questionnaires — Completion of questionnaires for the entire cohort:
  To assess hyperphagia and eating behaviour: BES, DEBQ and Hunger Score questionnaire To assess physical activity: short IPAQ To assess sleep behaviour: MCTQ To assess quality of life: EQ5D5L To assess digestive system disorders: GIQLI To assess anxiety and depression: HAD

SUMMARY:
The aim of the SEMASEARCH project is therefore to constitute a retrospective cohort, from the available data on patients already included in the ATUc/AP2, and prospective, on new patients who will initiate treatment according to the AP2 PUT, of 15 Specialized Obesity Centers in order to describe the effect of WEGOVY® treatment in this population. Thanks to a high phenotyping, subpopulations of interest will be identified to know the specifics of the effect of the treatment in these subgroups of interest. Secondary analyses will aim to look for clinical or biological biomarkers of success in the weight response to WEGOVY® in the entire prospective cohort, but also in specific subpopulations.

In summary, the analysis of the entire SEMASEARCH cohort and sub-populations of interest will be based on a complete clinical phenotyping of patients (included in retrospective and prospective studies), completed by ad hoc questionnaires and associated with biological markers (prospective) partly collected within the framework of the WEGOVY® AP (glycaemia, hepatic assessment, lipid assessment ) and partly from a biobank to test specific hypotheses (predictive role of leptin sensitivity, insulin sensitivity level, plasma level of endocannabinoids, etc.).

In addition, approaches using artificial intelligence (AI), notably machine learning, will make it possible to determine the variables or combination of variables that are most predictive of the weight response to treatment with WEGOVY® in the largest population. Indeed, individual weight loss in response to weight loss strategies is highly variable, whether purely related to lifestyle changes or pharmacological. Well-known factors associated with the ability to lose weight include adherence to lifestyle change, gender, age and specific medications. However, after controlling for these factors, differences in weight loss appear to persist in response to different interventions including pharmacological ones. Adaptation to energy deficit involves complex feedback mechanisms, and inter-individual differences are likely to arise from a range of poorly defined factors. Thus, a better understanding of the factors involved in inter-individual variability in response to WEGOVY® will help guide more personalised approaches to the management of these patients. AI techniques will be used to determine which combination of clinical or biological variables are most predictive of weight response.

ELIGIBILITY:
* Inclusion Criteria Male or female

Aged over 18 years

Patient included in the WEGOVY® ATU/AP program in one of the 14 participating CSOs: initial Body Mass Index (BMI) ≥ 40 kg/m² (Class III or morbid obesity) and presence of at least one weight-related comorbidity: treated hypertension, treated dyslipidemia, established cardiovascular disease, treated sleep apnea syndrome; and in the absence of therapeutic alternatives

Patient has been informed and has not objected to participation in the study

Patient affiliated with a French social security scheme

* Tagging Criteria to Identify Subpopulations of Interest (for classification purposes only - not a condition for inclusion)

  *1 Patients with a history of bariatric surgery:
  1. At least 1 year post-bariatric surgery (definitive technique or gastric band still in place)
  2. Defined as failure if:

     Initial %EWL < 50% (even without weight regain) and/or weight regain > 20% of lost weight compared to postoperative nadir

     *2 Patients with Binge Eating Disorder (BED):

     Defined by the clinician according to DSM-5 criteria for BED:

  a. Recurrent episodes of binge eating, characterized by both: Eating, in a discrete period of time, an amount of food that is definitely larger than what most individuals would eat in a similar time under similar circumstances A sense of lack of control over eating during the episode

  b. The binge eating episodes are associated with three (or more) of the following: Eating much more rapidly than normal Eating until uncomfortably full Eating large amounts of food when not physically hungry Eating alone due to embarrassment Feeling disgusted with oneself, depressed or guilty afterward

  c. Marked distress regarding binge eating

  d. The binge eating occurs, on average, at least once a week for 5 months

  e. The behavior is not associated with regular inappropriate compensatory behavior (e.g., purging, fasting, excessive exercise) and does not occur exclusively during anorexia nervosa or bulimia nervosa

  *3 Patients with rare monogenic or syndromic obesity: According to the French national guidelines (PNDS) for rare obesity causes: HAS website
  1. Includes:

     Hypothalamic (lesional) obesity, such as craniopharyngioma Genetic forms of obesity
  2. Most frequently encountered syndromes:

     Prader-Willi syndrome Bardet-Biedl syndrome 16p11.2 deletion or SH2B1 variant LEPR, POMC, PCSK1, and MC4R variants
     * 4 Older patients:

  <!-- -->

  1. Age > 60 years

     * 5 Patients with extreme obesity:

  a. BMI ≥ 60 kg/m²

  *6 Patients with obesity under psychotropic treatment:

Presence of one or more of the following treatments at baseline:

i. Antidepressants: Agomelatine, Amitriptyline, Citalopram, Clomipramine, Duloxetine, Escitalopram, Fluoxetine, Fluvoxamine, Imipramine, Iproniazid, Mianserin, Milnacipran, Mirtazapine, Moclobemide, Paroxetine, Sertraline, Tianeptine, Venlafaxine, Vortioxetine

ii. Antipsychotics: Amisulpride, Aripiprazole, Chlorpromazine, Clozapine, Cyamemazine, Flupenthixol, Fluphenazine, Haloperidol, Levomepromazine, Loxapine, Olanzapine, Pimozide, Pipamperone, Prochlorperazine, Quetiapine, Risperidone/Paliperidone, Sulpiride, Tiapride, Zuclopenthixol

iii. Mood stabilizers: Lithium carbonate, Carbamazepine, Lamotrigine, Oxcarbazepine, Sodium divalproate, Valpromide

iv. Psychostimulants: Methylphenidate

v. Anxiolytics: Antihistamines, anticonvulsants, or other anxiolytic agents

*7 Non-specific patients: Patients not meeting any of the above subpopulation criteria

- Exclusion Criteria

Pregnant or breastfeeding women

Persons under legal protection or guardianship

- Criteria for Early Study Withdrawal

Early withdrawal from the study will occur in the following cases:

The patient withdraws their non-opposition to participation

The patient discontinues treatment with WEGOVY® prematurely

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients included in the 15 centers in the indication of AP2 : Adults with an initial body mass index ≥ 40 kg/m2 (class III obesity or morbid obesity) in the presence of at least one treated comorbidity (treated hypertension, treated dyslipidemia, treated OSAS, established CVD) and included in the ATUc/AP2 WEGOVY®.
Sampling Method: Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Weight trends in patients included in the SEMASEARCH cohort at initiation and 12 months of treatment with WEGOVY®. | At initiation of treatment and 12 month of treatment
  Weight change between treatment initiation and 12 months after (greater than or equal to 10%)

SECONDARY OUTCOMES:
Proportion of responders at Month 12 | 12 months
  Defined as an absolute weight loss ≥10% from baseline to 12 months after treatment initiation
Change in binge eating and eating behavior | baseline, 6 and 12 months
  Change in binge eating and eating behavior based on Binge Eating Scale (BES)
  BES (Binge Eating Scale): 16-item self-report questionnaire, total score ranges from 0 to 46. Higher scores indicate more severe binge eating symptoms.
Change in sleep behavior based on Munich ChronoType Questionnaire (MCTQ) | baseline, 6 and 12 months
  Munich ChronoType Questionnaire (MCTQ) assesses sleep duration and chronotype using 6 questions. Derived variables include average sleep duration and midpoint of sleep. Higher sleep duration values reflect longer average sleep; midpoint values indicate chronotype.
Change in quality of life | baseline, 6 and 12 months
  EQ-5D-5L measures 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each rated on 5 levels. Results include:
  Index value: ranges from <0 (worse than death) to 1 (perfect health).
  Visual Analog Scale (VAS): 0-100, higher scores = better perceived health.
Change in physical activity based on the International Physical Activity Questionnaire - Short Form (IPAQ-SF) | baseline, 6 and 12 months
  The short version of the IPAQ (International Physical Activity Questionnaire) assesses overall physical activity and sedentary behavior over the past seven days. The questionnaire focuses on vigorous and moderate physical activity, walking, and time spent sitting (sedentary behavior), whether during leisure activities, work, daily life, or transportation. This short form includes 7 questions that can be self-administered or answered, for example, over the phone. The questionnaire categorizes individuals into three levels of activity: low, moderate, or high.
Change in gastrointestinal symptoms based on the reduced Gastrointestinal Quality of Life Index (GIQLI) | baseline, 6 and 12 months
  Reduced GIQLI has 13 items, each scored from 0 to 4. Total score ranges from 0 to 52. Higher scores indicate better gastrointestinal quality of life.
Change in anxiety and depression based on Hospital Anxiety and Depression Scale (HADS) | baseline, 6 and 12 months
  HADS has 14 items (7 for anxiety, 7 for depression). Each item is scored 0-3; subscale scores range from 0 to 21. Higher scores indicate more severe symptoms.
Evolution of metabolic comorbidities - Change in fasting glucose level (mg/dL) | baseline, 6 and 12 months
  Fasting plasma glucose will be collected from clinical records at each time point. Values are expressed in milligrams per deciliter (mg/dL). A decrease in glucose level reflects an improvement in glycemic control.
Number of participants with treatment-related adverse events reported in the eCRF at 6 and 12 months | 6 and 12 months
  All adverse events recorded in the electronic Case Report Form (eCRF) will be reported, classified by type, severity, and relationship to treatment.
Change in body composition - Change in fat mass percentage measured by Dual-Energy X-ray Absorptiometry (DXA) | baseline, 6 and 12 months
  Body fat percentage will be measured using DXA (dual-energy X-ray absorptiometry). Values are expressed as a percentage (%) of total body mass. A lower fat mass percentage over time is considered a positive outcome reflecting improved body composition.
Change in muscle strength based on chair stand test | baseline, 6 and 12 months
  Chair Stand Test: number of stands in 30 seconds.
Difference in lean mass between sarcopenic and non-sarcopenic patients | baseline, 6 and 12 months
  Lean body mass will be measured using Dual-Energy X-ray Absorptiometry (DXA) and/or Bioelectrical Impedance Analysis (BIA). Values will be expressed in kilograms (kg) and/or as a percentage of total body mass (%). The outcome will compare mean values between participants classified as sarcopenic and those classified as non-sarcopenic at each time point. Higher lean mass indicates better muscle preservation.
Change in body weight in each subpopulation | baseline, 6 and 12 months
  Body weight change from baseline to 6 and 12 months in subgroups of interest (e.g. BED, extreme obesity, sarcopenia, psychotropics)
Proportion of responders by subpopulation at Month 12 | baseline and 12 months
  Proportion of patients achieving ≥10% weight loss at 12 months in each subpopulation
Change in binge eating disorder symptoms in binge eating disorder subgroup | baseline and 12 months
  Change in binge eating disorder symptoms according to medical routine monitoring.
Change in prevalence of extreme obesity | baseline and 12 months
  Percentage of patients with BMI ≥60 kg/m^2 at baseline and at 12 months in extreme obesity subgroup
Change in psychotropic medication use at 12 months in patients on psychotropic medication | baseline and 12 months
  Proportion of patients who reduced, maintained, or increased psychotropic medication use.
Evolution of metabolic comorbidities - Change in liver enzymes (ALT and AST - U/L) | Baseline, 6 months, and 12 months
  Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels will be assessed as indicators of liver function. Values will be expressed in units per liter (U/L). Lower levels over time may reflect improved hepatic function or reduced liver inflammation.
Evolution of metabolic comorbidities - Change in lipid profile (total cholesterol, HDL, LDL, triglycerides - mg/dL) | Baseline, 6 months, and 12 months
  Lipid parameters will be collected from routine blood tests
Change in body composition - Change in lean body mass measured by Bioelectrical Impedance Analysis (BIA) | Baseline, 6 months, and 12 months
  Lean body mass will be assessed using bioelectrical impedance analysis (BIA). Results are expressed in kilograms (kg). An increase in lean mass over time indicates improved muscular composition and overall body health.
Difference in muscle strength between sarcopenic and non-sarcopenic patients | Baseline, 6 months, and 12 months
  Muscle strength will be assessed using Chair stand test measuring the number of repetitions in 30 seconds.
Change in eating behavior based on Dutch Eating Behavior Questionnaire (DEBQ) | Baseline, 6 months, 12 months
  DEBQ is a 34-item questionnaire assessing emotional eating, external eating, and cognitive restraint. Higher scores indicate more disordered eating patterns.
Change in hunger based on Hunger Score | Baseline, 6 months, 12 months
  Hunger Score consists of 4 items scored from 0 to 10. Higher score reflects greater hunger.

OTHER OUTCOMES:
Exploratory: Identification of clinical, behavioral, and biological predictors of response using interpretable machine learning models | Through study completion (up to 12 months after treatment initiation)
  Supervised machine learning algorithms will be used to identify predictive patterns for ≥10% weight loss response, based on clinical, behavioral, and biomarker data.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel DISSE, Pr, Principal Investigator — Hospices Civils de Lyon / Service Nutrition Diabétologie Endocrinologie
Locations (14):
- France (14):
  - Service Endocrinologie Diabétologie Nutrition APHP - Hôpital Jean Verdier, Bondy
  - Service de chirurgie APHP - GHU Nord Hôpital Louis Mourier, Colombes
  - Espace Médical Nutrition & Obésité (EMNO) Maison Médicale Valmy, Dijon
  - Service Endocrinologie Diabétologie Maladies Métaboliques CHU François Mitterrand Dijon, Dijon
  - Service Endocrinologie Diabétologie CHU de Grenoble, La Tronche
  - Service Endocrinologie Hôpital Conception - APHM, Marseille
  - Service Endocrinologie Diabétologie Nutrition Hôpital Lapeyronie - CHU Montpellier, Montpellier
  - Service Endocrinologie Diabétologie Nutrition CHU de Nantes - Hôpital Guillaume & René Laennec, Nantes
  - Service Nutrition APHP - GHU Pitié Salpêtrière, Paris
  - Service Nutrition Diabétologie Endocrinologie APHP - Hôpital Européen Georges-Pompidou (HEGP), Paris
  - Service Endocrinologie Hôpital Haut Léveque - CHU Bordeaux, Pessac
  - Service Endocrinologie Diabétologie Nutrition CHU Poitiers, Poitiers
  - Service Endocrinologie, Maladies Métaboliques et Nutrition Hôpital Rangueil (CHU Toulouse), Toulouse
  - Service Endocrinologie Diabète Nutrition Hôpitaux de Brabois - CHU Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Undecided